CLINICAL TRIAL: NCT03603522
Title: A Double-Blind Randomized Placebo Controlled Trial Investigating the Effects of DSM17938 on Capsaicin Evoked Coughs
Brief Title: Probiotics and Capsaicin Evoked Coughs
Acronym: PCEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: McMaster- DSM17938-5095
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2019-03

CONDITIONS: Atopic Asthma
Keywords: Cough; Capsaicin; Probiotics; TRPV1
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Participants will have a screening period followed by 28 days treatment with BioGaia DSM17938 or placebo, followed by a washout period and will then crossover to the opposite treatment received in the first part of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BioGaia-DSM17938 then Placebo Comparator (Experimental): 28 days treatment with BioGaia-DSM17938, followed by 28 days washout and then crossover to 28 days placebo comparator treatment.
  Interventions: Dietary Supplement: BioGaia-DSM17938; Other: Placebo Comparator: Placebo Control
- Placebo Comparator then BioGaia DSM17938 (Placebo Comparator): 28 days treatment with placebo comparator treatment, followed by 28 days washout and then crossover to 28 days treatment with BioGaia DSM17938.
  Interventions: Dietary Supplement: BioGaia-DSM17938; Other: Placebo Comparator: Placebo Control

INTERVENTIONS:
Dietary Supplement: BioGaia-DSM17938 — 2mL per day (1x10^9 CFU) per day taken orally for 28 days
Other: Placebo Comparator: Placebo Control — 2mL per day of placebo formulation taken orally for 28 days

SUMMARY:
Cough in asthma is a very common and troublesome symptom in asthma, which predicts severity and poor prognosis. Previous studies have shown that asthmatics have an exaggerated cough response to capsaicin. Currently available asthma treatment is not designed to target the cough reflex directly, so this presents an unmet need for patients. The treatment being tested in this study is the commercially available over the counter oral probiotic BioGaia® DSM17938. Based on clinical and pre-clinical evidence, it is hypothesized that TRPV1 antagonism with BioGaia® DSM17938 will result in a reduction in capsaicin evoked coughs in patients with asthma.

DETAILED DESCRIPTION:
Visit 1: Baseline Screening and Beginning of Treatment Period 1 Subjects will undergo consent, complete history, physical examination, spirometry, capsaicin cough challenge, skin prick testing (allergen and histamine), methacholine challenge, induced sputum and blood sampling. Eligible subjects will then be randomized with matched oral BioGaia DSM17938 and placebo and will be given for the next 4 weeks.

Visit 2: End of Treatment Period 1 Subjects will undergo spirometry, capsaicin cough challenge, skin prick testing, methacholine challenge, sputum induction and blood testing.

Washout: 28 day washout period prior to Visit 3.

Visit 3: Beginning of Treatment Period 2 Subjects wills undergo all the same tests performed in visit 2. Drug/Placebo will be given for the next 28 days.

Visit 4: End of Treatment Period 2 Subjects will undergo all the same tests performed in visit 2.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18
2. Able to understand and give written informed consent
3. Has a diagnosis of atopic asthma (based on at least one positive skin prick test and Methacholine PC20 ≤16 mg/ml)
4. FEV1 (forced expiratory volume at 1 second) ≥ 70% of predicted
5. Demonstrate a cough response to capsaicin

Exclusion Criteria:

1. Subjects who are in a pollen season that affects their asthma
2. Subjects who bronchoconstrict by more than 10% at the end of the full dose capsaicin cough challenge (assess after visit 1)
3. Subjects who do not display evidence of airway hyper-responsiveness (PC20>16mg/ml) (assess after visit 1)
4. Symptoms of upper respiratory tract infection (URTI) in the last 1 month which have not resolved.
5. Lower respiratory tract infection or pneumonia in the last 6 weeks.
6. Current smoker or ex-smoker with ≥10 pack year smoking history and abstinence of ≤6 months
7. Asthma exacerbation in the previous month requiring an increase or start of an ICS (inhaled corticosteroids) or OCS (oral corticosteroids)
8. Any asthma medication with the exception of infrequent (less than twice weekly) short-acting beta-agonist.
9. Subjects who have changed asthma medication within the past 4 weeks prior to screening
10. A previous asthma exacerbation requiring Intensive Care Unit (ICU) admission.
11. Significant other primary pulmonary disorders in particularly; pulmonary embolism, pulmonary hypertension, interstitial lung disease, lung cancer, cystic fibrosis, emphysema or bronchiectasis.
12. Pregnancy or breast-feeding
13. Use of ACE (angiotensin converting enzyme) inhibitors
14. Any centrally acting medication which in the view of the investigator could alter the sensitivity of the cough reflex
15. History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Emax | Day 1, Day 30, Day 59 and Day 89
  The maximum number of capsaicin evoked coughs

SECONDARY OUTCOMES:
ED50 (median effective dose) | Day 1, Day 30, Day 59 and Day 89
  The dose of capsaicin that evokes at least half the maximum number of coughs
Dose response | Day 1, Day 30, Day 59 and Day 89
  Changes in the capsaicin full dose response curves
C2 and C5 | Day 1, Day 30, Day 59 and Day 89
  Changes in the dose of capsaicin causing 2 coughs (C2) and 5 coughs (C5)
Responses to histamine | Day 1, Day 30, Day 59 and Day 89
  The wheal responses to graded doses of histamine skin prick testing
Itch Intensity | Day 1, Day 30, Day 59 and Day 89
  The intensity of itch after skin prick testing using a modified Borg scale (0-10)
T-Cell Cytokine | Day 1, Day 30, Day 59 and Day 89
  Inhibition of T-Cell cytokine responses to stimulation in blood
Sputum differential cell counts | Day 1, Day 30, Day 59 and Day 89
  Changes in sputum differential cell counts
PC20 | Day 1, Day 30. Day 59 and Day 89
  Changes in methacholine PC20

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Satia I, Cusack R, Stevens C, Schlatman A, Wattie J, Mian F, Killian KJ, O'Byrne PM, Bienenstock J, Forsythe P, Gauvreau GM. Limosilactobacillus reuteri DSM-17938 for preventing cough in adults with mild allergic asthma: A double-blind randomized placebo-controlled cross-over study. Clin Exp Allergy. 2021 Sep;51(9):1133-1143. doi: 10.1111/cea.13976. Epub 2021 Jul 8. PMID 34192396